CLINICAL TRIAL: NCT06054711
Title: Joint Aspiration in Dysfunctional Hip, Knee or Shoulder Prostheses (Chronic Infection or Implant Failure) "JAD-Pro"
Brief Title: Joint Aspiration in Dysfunctional Hip, Knee or Shoulder Prostheses
Acronym: JAD-Pro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Principal Investigator, SMARMOR, Director, Groupe Hospitalier Diaconesses Croix Saint-Simon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A00466-33
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Joint Prosthesis; Complications
MeSH Terms: interventions — Arthrocentesis

STUDY DESIGN:
Intervention Model Description: Prospective cohorte study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Joint Fluid Aspiration (Other): all included patients reporting prothesis complication will undergo a joint fluid aspiration
  Interventions: Other: joint puncture

INTERVENTIONS:
Other: joint puncture — Patients reporting complications such as pain hindering mobility or affecting quality of life, or any other symptoms suspecting prosthesis failure or infection will undergo joint fluid aspiration.

SUMMARY:
After a hip, knee or shoulder arthroplasty, the evolution is not always favorable. It can be marked by an infectious or non-infectious complication, most often implant failure. In this context, joint fluid aspiration (JFA) is indicated to document a prosthetic joint infection (PJI) or to bring to light arguments for implant failure. Nevertheless, opinions differ on its indication for microbiological identification. Some teams perform it systematically when faced with a prosthesis dysfunction. Others, only in the presence of suggestive signs of PJI. Finally, others never perform it.

Based on clinical, radiological and biological (CRP) signs, at the preoperative stage and before JFA, we classify our patients into 3 groups: supposedly septic (chronic joint infection), supposedly aseptic (implant failure) or intermediate (Unknown). This last group, often encountered in consultation, poses a diagnosis problem more than the others.

In our experience, JFA is an essential diagnosis tool in these 3 groups of patients. It helps to choose the surgical strategy. In addition, the dosage of biomarkers in the joint fluid as the alpha defensin, the leucocyte esterase and the CRP could provide an additional argument to investigate the infectious origin or not, in particular in difficult cases.

In summary, the disagreement on the usefulness of JFA in case of PJI suspicion and any other prosthetic dysfunction, the lack of data on large prospective studies and our questioning about the contribution of JFA in the aseptic and intermediate group of patients, motivated us to set up this study to evaluate the interest of the JFA for the preoperative diagnosis, as well as that of the dosage of biomarkers in the joint fluid.

DETAILED DESCRIPTION:
Visit V0: corresponds to the first consultation. After informing and obtaining the consent of the patient, the investigator will collect the anamnesis, clinical, radiological and biological data, then will indicate the anticipated medico-surgical strategy. The FJA will be prescribed during this consultation, as well as the dosage of the CRP in blood the same day as the FJA.

Then, the investigator will classify the patient (primary classification) in one of the three groups the groups: supposedly septic, supposedly aseptic or intermediate.

A reclassification of patients (secondary classification) will be done, based on the bacteriological results of the FJA (positive, negative and doubtful). Biomarker results will not be disclosed or considered for patient care.

Visit V1: corresponds to the day of the FJA in the x.ray department and the blood sample in the central laboratory for the CRP dosage.

During FJA, 2 ml of additional joint fluid will be collected in addition to the volume usually collected for CRP, Leukocyte Esterase and alpha defensin dosage in joint fluid. Alpha defensin dosage will be performed only in patients in the intermediate group with a negative FJA.

Visit V2: Day of prosthesis revision in the event of chronic PJI or mechanical prosthesis dysfunction (Implant failure) requiring surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient consent to participate in the study.
* Patient aged over 18 years
* Patient with hip, knee or shoulder joint prosthesis
* Patient who has the Indication to perform a FJA, whatever the cause of revision (mechanical, septic)
* Over one-month symptoms evolution for patients suspected of infection

Exclusion Criteria:

* Acute prosthesis infection with less than one-month symptoms' duration
* Antibiotic therapy between preoperative FJA and intraoperative samples
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-02-07 (Estimated); Study Completion 2024-08-07 (Estimated)

PRIMARY OUTCOMES:
Analysis of the bacteriological concordance between JFA and perioperative samples | From JFA till perioperative samples bacteriological analysis termination
  Number of patients whose JFA is concordant with that of the perioperative samples

CONTACTS AND LOCATIONS:
Overall Officials: Simon MARMOR, MD, Principal Investigator — Groupe Hospitalier Diaconesses Croix Saint-Simon
Locations (1):
- Groupe Hospitalier Diaconesses Croix saint Simon, Paris, France